CLINICAL TRIAL: NCT01465035
Title: A Phase I Study to Determine the Safety and Immunogenicity of Co-administration of the Candidate Influenza Vaccine MVA-NP+M1 and Seasonal Influenza Vaccine
Brief Title: A Study to Determine the Safety and Immunogenicity of Co-administration of the Candidate Influenza Vaccine MVA-NP+M1 and Seasonal Influenza Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Flu003
Record Dates: First submitted 2011-10-21; First posted 2011-11-04 (Estimated); Last update posted 2012-11-29 (Estimated); Status verified 2012-11

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TIV and MVA-NP+M1 (Experimental): Co-administration group
  1 dose of seasonal influenza vaccine (TIV) and 1 dose of 1.5 x108pfu MVA-NP+M1
  Interventions: Biological: TIV and MVA-NP+M1
- Saline placebo and seasonal influenza vaccine TIV (Placebo Comparator): Control group
  1 dose of seasonal influenza vaccine (TIV) and 1 dose of a saline placebo
  Interventions: Biological: Saline placebo and seasonal influenza vaccine TIV

INTERVENTIONS:
Biological: TIV and MVA-NP+M1 — 1.5 x 108 pfu MVA-NP+M1, intramuscular injection into the thigh. Inactivated Influenza Vaccine (Split Virion) 0.5ml (containing 15 micrograms of haemagglutinin, intramuscular injection into the thigh
  Arms: TIV and MVA-NP+M1
Biological: Saline placebo and seasonal influenza vaccine TIV — Saline placebo, intramuscular injection into the thigh. Inactivated Influenza Vaccine (Split Virion) 0.5ml (containing 15 micrograms of haemagglutinin, intramuscular injection into the thigh
  Arms: Saline placebo and seasonal influenza vaccine TIV

SUMMARY:
This is a single blinded placebo controlled phase I study, to assess the safety and immunogenicity of co-administration of the candidate influenza vaccine MVA-NP+M1 with seasonal influenza vaccine. All volunteers recruited will be adults aged 50 and over.

The rationale behind co-administration of MVA-NP+M1 with a seasonal influenza vaccine (TIV) is that the immune system will be stimulated to produce both influenza specific T cells and influenza specific antibodies.

ELIGIBILITY:
Inclusion Criteria:

Men and women aged 50 or over with no upper age limit

* Resident in or near Oxford for the duration of the vaccination study
* Able and willing (in the Investigators' opinions) to comply with all study requirements
* Willing to allow the investigators to discuss the volunteer's medical history with their General Practitioner
* For females who are not post-menopausal, a negative pregnancy test on the day of vaccination and agreement to practice effective contraception for the duration of the study
* Agreement to refrain from blood donation during the course of the study
* Written informed consent

Exclusion Criteria:

Participation in another research study involving an investigational product in the 30 days preceding enrolment, or planned use during the study period

* Receipt of MVA or smallpox vaccines in the last 5 years, or receipt of the 2011/12 seasonal influenza vaccine prior to entering the study.
* Administration of immunoglobulins and/or any blood products within the three months preceding the planned administration of the vaccine candidate
* Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months (inhaled/topical steroids are allowed)
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine, e.g. egg products
* Any history of anaphylaxis in reaction to vaccination
* Recent treatment for cancer (except basal cell carcinoma and cervical carcinoma in situ)
* History of serious psychiatric condition
* Suspected or known current injecting drug or alcohol abuse (as defined by an alcohol intake of greater than 42 units every week)
* Seropositive for hepatitis B surface (HBsAg) or hepatitis C virus (antibodies to HCV)
* For pre-menopausal females, pregnancy, lactation or willingness/intention to become pregnant during the study
* Any other significant disease, disorder or finding (including blood test results), which, in the opinion of the Investigators, would either put the volunteer at risk because of participation in the study, or may influence the result of the study.
* No response / confirmation from GP regarding previous medical history

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-10; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Safety of co-administration of MVA-NP+M1 and seasonal influenza vaccine. | Participants will be followed for the duration of the study, an expected average of 6 months
  The specific endpoints for safety and reactogenicity will be actively and passively collected data on adverse events.

SECONDARY OUTCOMES:
Immune response generated by co-administration of MVA-NP+M1 and seasonal influenza vaccine | Participants will be followed for the duration of the study, an expected average of 6 months
  To assess immune response generated by co-administration of MVA-NP+M1 by interferon-gamma ELISpot and ELISA.

CONTACTS AND LOCATIONS:
Overall Officials: Adrian VS Hill, DPhil FRCP, Principal Investigator — University of Oxford
Locations (1):
- Centre for Clinical Vaccinology and Tropical Medicine, Churchill Hospital, Oxford, United Kingdom